CLINICAL TRIAL: NCT05422963
Title: Multiple-Center Retrospective Study of Severe and Critical COVID-19 in Shanghai
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCCS-2022-1
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe and critical COVID-19: 1. hospital admission time more than 24 hours
  2. meet the standard of definition of severe and critical COVID-19 in "Diagnosis and Treatment Plan for new Coronavirus Pneumonia (Ninth Edition)"

SUMMARY:
This study is to clarify the clinical characteristics of severe and critical COVID-19 from March 1st ,2022 to June 9th, 2022 in Shanghai and to explore the relationship between the characteristics and prognosis in these patients.

DETAILED DESCRIPTION:
1. To Describe the clinical characteristics of severe and critical COVID-19.
2. To analyze the relationship between the clinical characteristics and their clinical prognosis;
3. To analyze the relationship between clinical intervention and their clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* severe and critical covid-19 patients who met the "Diagnosis and Treatment Plan for new Coronavirus Pneumonia (Ninth Edition)"
* admission time more than 24 hours

Exclusion Criteria:

* admission time less than 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: severe and critical COVID-19 patients admitted to specific medical systems in Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | one year
  28-day mortality of severe and critical COVID-19

SECONDARY OUTCOMES:
60-day mortality | one year
  60-day mortality of severe and critical COVID-19
ICU length of stay | one year
  ICU length of stay
the percentage of organ failure | one year
  the percentage of organ failure include respiratory，circulatory failure and so on
time for virus to turn negative | one year
  time for COVID-19 from positive to negative
The overall description | one year
  The overall description of the clinical characteristics in severe and critical covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Erzhen Chen, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
the data are not publicly available due to the privacy and ethical restriction.